CLINICAL TRIAL: NCT03099798
Title: Traumatic Splenic Injury and Management (SPLENIQ Study) Quality of Life and Clinical Outcomes of Treatment for Splenic Injury After Trauma
Brief Title: Traumatic Splenic Injury and Management (SPLENIQ Study)
Acronym: SPLENIQ
Status: Completed | Type: Observational
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: Erasmus Medical Center (Other); Maasstad Hospital (Other); Albert Schweitzer Hospital (Other); Amphia Hospital (Other); Tilburg University (Other); Leiden University Medical Center (Other); Amsterdam UMC, location VUmc (Other); Medisch Spectrum Twente (Other); Radboud University Medical Center (Other); Isala (Other)
Responsible Party: Sponsor
Other Study IDs: NL54542.028.16 / P1609
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life; Spleen Injury; Trauma; Splenic Artery Embolization
MeSH Terms: conditions — Wounds and Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-Operative Management (NOM)/Observational: Patients "treated" observationally for (traumatic) spleen injury.
  Interventions: Other: Questionnaires
- Splenic Artery Embolization: Patients treated with splenic artery embolization for (traumatic) spleen injury.
  Interventions: Other: Questionnaires; Diagnostic Test: MRI abdomen
- Surgery: Patients treated surgically for (traumatic) spleen injury.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — All patients will complete a number of questionnaires at different time points.
  * SF-12, WHOQoL-Bref, EQ-5D-5L, iPCQ, iMCQ
  * 1 week, 1 month, 3, 6 and 12 months after treatment
Diagnostic Test: MRI abdomen — Patients who were treated with splenic artery embolization will also undergo an MRI one month and one year after treatment.
  Groups: Splenic Artery Embolization

SUMMARY:
OBJECTIVE:

To determine the quality of life (QOL) and clinical outcome after conservative therapy, embolization (proximal versus distal) or surgery in patients with traumatic splenic injury. Secondary aims: (I) to examine therapy-related complications, (II) to establish the necessity of additional therapies, (III) the assessment of splenic function related to splenic morphology (MR imaging) after embolization and (IV) to find the prognostic factors for failure of non-operative management (NOM) in patients with splenic injuries. Finally, with the acquired data from this study a patient-oriented protocol will be provided for the management of traumatic splenic injury.

HYPOTHESIS:

The investigators expect that NOM is superior to surgery with regard to QOL, clinical outcome and splenic function. Embolization will need more additional therapies. Splenic morphology is related to splenic immune function. Expected prognostic factors are age above 40, ISS >25 and a splenic injury grade of 3 or higher.

STUDY DESIGN:

A combination of a retrospective and a prospective multicentre cohort study. This protocol involves the prospective part of the study.

STUDY POPULATION/DATASET:

Patients who enter the participating hospitals between March 2017 and December 2018 with splenic injury will be asked to participate. The follow-up period will be one year with regard to QOL, clinical symptoms and imaging.

INTERVENTION:

All patients will complete a number of questionnaires at different time points. The patients who were treated with splenic artery embolization (SAE) will undergo an MRI one month and one year after treatment.

OUTCOME MEASURES:

Primary outcome is QOL. Secondary outcomes are clinical symptoms and imaging.

SAMPLE SIZE:

Approximately 100 patients will be included per year during the inclusion phase.

DATA ANALYSIS:

With regard to the prospective data linear modelling will be performed.

COLLABORATION/CONNECTION:

Tilburg University, Erasmus Medical Center Rotterdam, Maasstad Hospital Rotterdam, Albert Schweitzer Hospital Dordrecht, Amphia hospital Breda, Leiden University Medical Center, VU University Medical Center Amsterdam, Medical Spectrum Twente, Radboud University Nijmegen, Isala Zwolle.

TIME SCHEDULE:

Year 1: literature search and conducting the retrospective study and analyses. Years 1-3: inclusion prospective study and follow-up of patients. Year 4: finishing follow-up data collection and analysing.

ELIGIBILITY:
Inclusion Criteria:

* Splenic injury after blunt abdominal trauma (confirmed by FAST and/or CT)
* The patient underwent NOM/SAE/splenectomy for the management of traumatic splenic injury
* The treatment took place in the period from March 2017 to December 2018 at one of the five selected hospitals
* 18 years or older.

Exclusion Criteria:

* Insufficient knowledge of the Dutch language
* Patients who died during or after treatment are (of course) excluded for questionnaires and MRI, not for clinical outcomes

Exclusion for MRI only:

- Patients treated with SAE: patients who do not want to or are not able to undergo an MRI abdomen (for example pregnant women or other contraindications for MRI). Patients excluded for MRI still need to fill out the questionnaires. Also, their clinical outcomes will be processed in the database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with splenic injury after blunt abdominal trauma confirmed by ultrasound (US/FAST) and/or computed tomography (CT) at the primary trauma screening at the 5 selected hospitals between March 2017 and December 2018 will be asked to participate in this study as soon as they can talk and are lucid. Patients receive a verbal and written explanation about the study. The time for consideration is one week. When a patient is willing to participate he/she will be asked to sign a consent form. When patients agree to participate, they are included for follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life: baseline (within 1 week after treatment) | One week after treatment
  WHOQoL-Bref questionnaire, SF-12 and EQ-5D-5L questionnaires
Quality of life: 1 month follow-up | One month after treatment
  WHOQoL-Bref questionnaire
Quality of life: 3 months follow-up | Three months after treatment
  WHOQoL-Bref questionnaire
Quality of life: 6 months follow-up | Six months after treatment
  WHOQoL-Bref questionnaire
Quality of life: one year follow-up | One year after treatment
  WHOQoL-Bref questionnaire
Change in health status: SF-12 | One week, 1 month and 3, 6 and 12 months after treatment
  SF-12 questionnaire
Change in health related quality of life: EQ-5D-5L | One week, 1 month and 3, 6 and 12 months after treatment
  EQ-5D-5L questionnaire

SECONDARY OUTCOMES:
Clinical Outcome | One year follow-up
  Data obtained from the patient records (e.g. complications, need for re-intervention, hospital stay, return to daily activities)
Cost-effectiveness | One year follow-up
  The overall cost-effectiveness will be assessed with the iPCQ and iMCQ questionnaires, completed at different time points
Imaging Outcome after Embolization (one month after treatment) | One month after embolization
  Splenic morphological characteristics (e.g. volume, necrosis, splenosis, calcifications or chronic infarction morphology)
Imaging Outcome after Embolization (one year after treatment) | One year after embolization
  Splenic morphological characteristics (e.g.volume, necrosis, splenosis, calcifications or chronic infarction morphology)
Splenic Artery Embolization characteristics | One year follow-up
  Difference between proximal versus distal embolization
Prognostic factors for failure of Non-Operative Management | One year follow-up
  A recent study suggests that there are prognostic factors for failure of NOM in the treatment of adults with (blunt) splenic injury. Strong evidence exists for: age of 40 years or above, Injury Severity Score (ISS) of 25 or greater and American Association for the Surgery of Trauma (AAST) splenic injury grade of 3 or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanda de Vries, Prof. dr., Principal Investigator — Project leader (ETZ Tilburg, Tilburg University)
Locations (10):
- Netherlands (10):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Amphia Hospital, Breda, North Brabant
  - Elisabeth-Twee Steden Hospital, Tilburg, North Brabant
  - VU University Medical Center, Amsterdam, North Holland
  - Medical Spectrum Twente, Enschede, Overijssel
  - Isala, Zwolle, Overijssel
  - Albert Schweitzer Hospital, Dordrecht, South Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Maasstad Hospital, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raaijmakers CP, Lohle PN, Lodder P, de Vries J. Quality of Life and Clinical Outcome After Traumatic Spleen Injury (SPLENIQ Study): Protocol for an Observational Retrospective and Prospective Cohort Study. JMIR Res Protoc. 2019 Apr 26;8(5):e12391. doi: 10.2196/12391. PMID 31066709
- See also: Related Info — https://www.zonmw.nl/nl/onderzoek-resultaten/kwaliteit-van-zorg/programmas/project-detail/topzorg/traumatic-splenic-injury-and-management/
- See also: Related Info — https://www.etz.nl/TopZorg/Behandeling-traumatisch-miltletsel